CLINICAL TRIAL: NCT05326334
Title: THERApeutic Outcomes Related to Gut microBIOME in Glioblastoma (GBM) Patients Receiving Chemo-radiation: A Prospective Observational Study
Brief Title: THERApeutic Outcomes Related to Gut microBIOME in Glioblastoma (GBM) Patients Receiving Chemo-radiation (THERABIOME-GBM)
Acronym: THERABIOME-GBM
Status: Recruiting | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 3603
Record Dates: First submitted 2022-03-02; First posted 2022-04-13 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Glioblastoma, IDH-wildtype
Keywords: Gut microbiome; Glioblastoma multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This study collects patient stool samples for 16S RNA analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a pilot or feasibility study to test the study plan and to find out whether enough participants will join a larger study and accept the study procedures. Eligible participants (adults with newly diagnosed glioblastoma multiforme [GBM] and had a good tumour resection [>= 70% of initial tumour volume] and plan to receive 6 weeks of chemoradiation followed by up to 6 months of chemotherapy) are asked to donate their own stool samples at 4 different time points during their treatment course. Participants will also complete a 7-day diet diary and two questionnaires about their health-related quality of life.

Glioblastoma multiforme (GBM) is the most common and aggressive form of primary brain cancer in adults. The current best evidence-proven treatment for GBM includes maximum safe tumour resection, brain radiation over a 6-week period given with chemotherapy pills called temozolomide (Brand name: Temodal or Temodar), followed by approximately 6 months / cycles of temozolomide. Despite these treatments, the average life expectancy is generally less than 2 years.

Researchers are recognizing that the immune system has an important role in directing the effectiveness of chemotherapy, radiation, and newer therapies such as immunotherapies. Some immunotherapies have been quite successful in improving cancer control and survival in other cancers like melanoma (an aggressive skin cancer), but when these drugs were given to patients with GBM, there appeared to only be a small effect. Therefore, finding ways to make existing and new treatments work better should be a priority. Recent scientific studies have shown that the bacteria that make up our stool, often referred to as the gut microbiome, play a major role in regulating the immune system. For example, researchers were able to make patients with melanoma who previously did not respond to immunotherapy become responsive to the treatment after receiving a stool transplant from responders to immunotherapy. This provides proof of concept that we could modify the body's immune environment to favour cancer killing by changing a person's gut bacteria environment.

The role of the gut bacteria in patients with brain cancer is poorly understood as very few studies have been published about it in this population. We believe that understanding the composition of the gut microbiome and how it relates to the effectiveness and side effects of treatments in GBM patients will be an important first step to understanding how we can modify the gut microbiome to improve outcomes for patients living with GBM.

DETAILED DESCRIPTION:
This is a prospective observational study designed to assess changes in the gut microbial composition and diversity in prospectively collected stool samples at important time points throughout GBM treatment and surveillance and to correlate that with patient survival outcomes and radiation necrosis.

Objectives:

1. To assess feasibility of stool sample collection, banking, and analysis throughout the treatment course of GBM patients.
2. To determine the association of gut microbiome composition with survival outcomes in isocitrate dehydrogenase (IDH) type 1 wild type glioblastoma multiforme (GBM)
3. To assess the association of gut microbiome composition with radiation necrosis

Hypothesis: We hypothesize that stool collection and microbiome analysis taken from the time of diagnosis to disease recurrence will be feasible in Ottawa. Secondly, we hypothesize that in patients with newly diagnosed World Health Organization (WHO) Grade 4, IDH-1 R132H (Arginine to histidine mutation at site 132) wild-type glioblastoma (GBM) receiving chemoradiation (Stupp regimen), increased microbial diversity and abundance of microbiota found to be favorable in other cancers will have better survival outcomes compared to decreased gut microbial diversity and relative abundance of microbiota found to be unfavorable in other cancers

Study sample size: n=20.

This study aims to enroll a prognostically uniform population presenting with newly diagnosed GBM at a single cancer center. The primary aim of the study is to establish feasibility of conducting such a study in Ottawa.

Primary Outcome(s) The primary outcome is study feasibility. Feasibility will be determined by the following co-primary endpoints.

1. Stool sample obtained at pre-radiation, post-radiation (pre-adjuvant temozolomide chemotherapy), and at time of disease relapse in ≥ 70% of enrolled patients
2. Complete 15-patient (75% of target sample size) enrollment within 2 years
3. Stool sample volume and quality sufficient for analysis in ≥ 75% of collected samples

Secondary Outcomes

1. Overall survival (OS) and progression-free survival (PFS) in pre-defined subgroups with high gut microbial diversity and relative abundance of taxa associated with favorable outcomes in other cancers vs. low diversity and unfavorable taxa subgroup.
2. Gut microbial taxonomy and diversity (i.e., microbiome make up) in late progressors versus early progressors
3. Differences in gut microbiome in patients with and without post-radiation necrosis.

Timing of Standard of Care Visits and Study Procedures

Participants will be followed as part of standard of care, which involves visits at the following time points:

* Baseline: post-surgery but before temozolomide (chemo) plus radiation (pre-chemoRT)
* 3-month: approximately one month after 6 weeks of chemoradiation (post-chemoRT), but before starting maintenance phase of chemotherapy
* Months 4 to 9: monthly while on maintenance phase of chemotherapy
* Every 2-3 months after completing maintenance chemo, usually corresponding to MRI scans

There are 4-5 time points during which study participants will be asked to participate in study procedures

1. Stool sample collection - 4 time points from the time of enrollment

   * Baseline - pre-chemoRT
   * 3 month - post-chemoRT
   * 1 to 3 months after completing maintenance chemotherapy. As a result, this time point may vary (e.g., could be at 9-month mark if they finished 6 cycles of maintenance chemotherapy on schedule, but may be earlier or later, if patients stop maintenance chemo early or treatments repeatedly get delayed).
   * Disease recurrence (12-week window of confirmed recurrence date)
2. 7-day diet diary - 4 time points from time of enrollment.

   * Baseline: pre-chemoRT
   * 3-month: post-chemoRT
   * 9-month: usually corresponds to after maintenance chemo
   * 12 month: even further out from completion of chemo
3. European Organization for Research and Treatment of Cancer (EORTC)-quality of life questionnaire (QLQ)-C30 and EORTC-QLQ-BN20 questionnaires - 5 time points from time of enrollment

   * Baseline: pre-chemoRT
   * 3-month: post-chemoRT
   * 6-month: usually mid-maintenance chemo
   * 9-month: usually corresponds to after maintenance chemo
   * 12-month: even further out from completion of chemo

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed WHO grade 4 glioblastoma, IDH-1 R132H wild type
* Maximum safe resection (≥70% of initial tumor volume resected)
* Age ≥ 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 or ECOG 2 if on ≤ 8 mg/day of dexamethasone (or bioequivalent)
* Plan to receive 60 Gy / 30 fractions of radiation with temozolomide within 12 weeks of surgery
* Patient or substitute decision maker able to provide written informed consent

Exclusion Criteria:

* Metastatic cancer or secondary cancer that could affect interpretation of primary and secondary study outcomes
* Receiving additional systemic therapy / clinical intervention for glioblastoma that would prevent a uniform treatment cohort with temozolomide and radiation x 6 weeks followed by adjuvant temozolomide 150-200 mg/m2 on days 1-5 every 28 days for up to 6 cycles.*
* Inability to collect study stool samples
* Any diagnosis or medical condition, physical and / or psychological, that the investigator feels precludes the patient from participation in the study.

  * If there is a new standard of care treatment for newly diagnosed GBM before the first patient is enrolled (e.g., Optune Tumor Treating Fields), then we will allow all patients on this study to adopt the new standard of care therapy. To allow for maximum patient accrual, if patient chooses to enroll on an open label randomized therapeutic study whereby the control arm involves only the standard of care treatment, then patients enrolled in the control arm could be eligible for this study at the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IDH-1 R132H wild type WHO grade 4 glioblastoma multiforme is the most common type of primary brain cancer. This study enrolled prognostically similar patients (at least 70% tumour volume resection, ECOG PS 0-2, eligible to receive RT 60 Gy/30 fractions)
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility of collecting stool samples | 2 years
  Feasibility is met if stool samples obtained at pre-radiation, post-radiation (pre-adjuvant temozolomide chemotherapy), and at time of disease relapse in ≥ 70% of enrolled patients
Feasibility of participant enrollment | 2 years
  Feasibility is met if 15 participants (75% of target sample size) are enrolled within 2 years
Feasibility of stool sample analysis | 2 years
  Feasibility is met if 16S RNA analysis is feasible in ≥ 75% of collected stool samples

SECONDARY OUTCOMES:
Progression-free survival in favourable and unfavourable gut microbiota subgroups | 5 years
  Favourable and unfavourable gut microbiota subgroups will be pre-defined by gut microbial diversity (high vs. low) and relative abundance of taxa associated with favorable and unfavorable outcomes seen in other cancers
Gut microbial composition in late versus early progressors | 5 years
  Gut microbial taxonomy and diversity (i.e., microbiome make up) in late progressors versus early progressors
Gut microbial composition associated with radiation necrosis | 2 years
  Differences in gut microbiome in patients with and without post-radiation necrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No